CLINICAL TRIAL: NCT05138276
Title: Effect of Autologous Cord Blood Mononuclear Cells for Digestive System in Preterm Neonates
Acronym: ACBMNC
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Women and Children Hospital (Other)
Responsible Party: Principal Investigator, yang jie, Professor, Guangdong Women and Children Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Guangdong Women and Children H
Record Dates: First submitted 2021-05-21; First posted 2021-11-30 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Neonatal Necrotizing Enterocolitis; Growth and Development; Preterm Infants; Nutrition
Keywords: Necrotizing enterocolitis; Preterm infants; Prevention; cord blood mononuclear cells
MeSH Terms: conditions — Enterocolitis, Necrotizing | interventions — Sodium Chloride

STUDY DESIGN:
Masking Description: Triple (Participant, Care Provider, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autologous cord blood mononuclear cells (Experimental): Autologous Umbilical Cord Blood Mononuclear Cells Therapy 24 hours after birth ,dose is 50 million cells/kg
  Interventions: Other: Autologous Umbilical Cord Blood Mononuclear Cells Therapy
- Placebo (Placebo Comparator): 0.9% sodium chloride infusion 24 hours after birth
  Interventions: Drug: 0.9% Sodium Chloride

INTERVENTIONS:
Other: Autologous Umbilical Cord Blood Mononuclear Cells Therapy — Autologous Umbilical Cord Blood Mononuclear Cells Therapy in preterm for prevention of NEC
  Arms: Autologous cord blood mononuclear cells
Drug: 0.9% Sodium Chloride — 0.9% Sodium Chloride in control group
  Arms: Placebo

SUMMARY:
Pre-clinical animal studies provide robust evidence regarding the beneficial effect of stem cells for intestinal disease.

This single-center, randomized, controlled, blinded trial assessed the effect of a single intravenous infusion of autologous cord blood MNCs (ACBMNCs) in preventing NEC in preterm neonates,and influence on growth and development.

DETAILED DESCRIPTION:
Study design and settings:

This study will be a randomized, placebo-controlled, double-blinded, single-center trial. A total of 45 singleton preterm infants (GS<33 weeks) of fulfilling the eligibility criteria will be enrolled. According to the infusion of umbilical cord blood mononuclear cells and equal dose placebo, the premature infants were divided into infusion group and control group. The two groups were matched with gender, gestational age and birth weight as stratified variables and 1:2 (the gender was the same, and the difference between gestational age and birth weight was the smallest).

Trial treatment methods: Study design and settings:

This study will be a randomized, placebo-controlled, double-blinded, single-center trial. A total of 30 pairs of monozygotic twins fulfilling the eligibility criteria will be enrolled. Subsequently, one baby of each twin will be randomly divided into the ACBMNC infusion group or control (placebo) group.

Trial treatment methods:

Soon after the preterm infant was deliveried, written consent was signed by the parents, and autologous cord blood infusion was applied to the baby in addition to routine treatment. Those assigned to the ACBMNC group received an infusion of ACBMNC . Those in control group received an infusion of a placebo solution. Informed consent before birth is signed. Preterm infants in the ACBMNC infusion group will have their umbilical cord blood collected after birth, and then their umbilical cord blood will be separated through Guangdong Province umbilical cord blood Bank to obtain mesenchymal stem cells. Within 24h after birth, ACBMNC group received an infusion of mesenchymal stem cells timely, while control (placebo) group received an infusion of a placebo solution which is normal saline with the same volume. Cell dose for all patients was targeted at 5×107 cells per kilogram.

ELIGIBILITY:
Inclusion Criteria: (1) born at the study hospital; (2) singleton birth; (3) 26<GA <32 weeks; (4) free of severe congenital anomalies or genetic syndromes;

Exclusion criteria： (1) mothers with clinical chorioamnionitis; (2) the mother was opsitive for hepatitis B (HBsAg and/or HBeAg), hepatitis C (anti-HCV), syphilis, HIV (anti-HIV-1 and -2), and IgM against cytomegalovirus, rubella, toxoplasma, and herpes simplex viruses; (3) consent was not obtained from the parents or guardians; and (4) after processing, UCB cells were not available.

Ages: 26 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The occurrence of Necrotizing enterocolitis in hospitalization | up to one year
  NEC rate

SECONDARY OUTCOMES:
The severity of Necrotizing enterocolitis | up to one year
  severe NEC
The occurrence of feeding intolerance | up to one year
  Other outcomes
The occurrence of other intestinal disease | up to one year
  Other outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Jie Yang, PHD, Principal Investigator — Guangdong Women and Children Hospital
Locations (1):
- Jie Yang, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ballen KK, Gluckman E, Broxmeyer HE. Umbilical cord blood transplantation: the first 25 years and beyond. Blood. 2013 Jul 25;122(4):491-8. doi: 10.1182/blood-2013-02-453175. Epub 2013 May 14. PMID 23673863
- [Background] Mezey E, Nemeth K. Mesenchymal stem cells and infectious diseases: Smarter than drugs. Immunol Lett. 2015 Dec;168(2):208-14. doi: 10.1016/j.imlet.2015.05.020. Epub 2015 Jun 4. PMID 26051681